CLINICAL TRIAL: NCT07330427
Title: Impact of Health Education on Knowledge, Attitude and Practice of Post-exposure Prophylaxis Among Health Care Workers at Aswan University Hospital, Egypt
Brief Title: Impact of Health Education on Knowledge, Attitude and Practice of Post-exposure Prophylaxis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Fatma Ali Mahmoud Hussein, Demonstrator at Public Health and Community Medicine, Faculty of medicine, Aswan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Post-exposure prophylaxis
Record Dates: First submitted 2025-12-11; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-06

CONDITIONS: Post Exposure Prophylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Care workers (Experimental): About 340 participants of heath care workers undergoing assessment of knowledge, attitude and practice about post-exposure prophylaxis among health care workers at Aswan university hospital, Egypt Then they will undergo lecturers about about post-exposure prophylaxis, then reassessment will be done after 3 months
  Interventions: Procedure: Health Education

INTERVENTIONS:
Procedure: Health Education — 1. Assess the baseline knowledge, attitudes and practices of health care workers at Aswan university hospital towards postexposure prophylaxis against blood-borne viral infection.
  2. Provide an intense post exposure prophylaxis health education sessions.
  3. Evaluate changes in post exposure prophylaxis knowledge, attitudes and practices after the health education intervention.

SUMMARY:
Occupational exposure to blood-borne pathogens, such as human immune-deficiency virus (HIV), hepatitis B virus (HBV), and hepatitis C virus (HCV) for healthcare workers through contact with human blood and body fluids has become a major health concern as it poses a risk of transmission of these infectious agents.

According to the World Health Organization (WHO) report, about three million HCWs are exposed to blood-borne pathogens each year, of which 170,000 are exposed to HIV infections, 2 million to HBV infections, and 0.9 million to HCV infections. Most of the time, healthcare providers get exposure through the splash of blood or other body fluids into the eyes, nose, or mouth or nonintact skin exposure, and percutaneous injury occurs as a result of a break in the skin caused by a needlestick or sharps contaminated with blood or body fluids

DETAILED DESCRIPTION:
Post exposure prophylaxis is defined by the World Health Organization (WHO) as the medical intervention offered to prevent the transmission of blood-borne diseases following a potential exposure to HIV, HBV, HCV, and other viruses.

In developing regions, 40%-65% of HBV and HCV infections in health care workers are attributable to percutaneous occupational exposure .Approximately 3 out of 35 million HCWs worldwide experience needlestick injuries (NSIs) annually, exposing them to blood-borne pathogens .

In Egypt, like many developing countries, few efforts have been undertaken to raise awareness about needlestick injury (NSI) among HCWs . There is a lack of regulations and policies to protect HCWs from exposure. HCWs rarely receive training in infection control and standard precautions, even though these are low-cost solutions to reducing the risk of sharp injuries and have a high likelihood of being adopted .

There is a lack of data and surveillance concerning health care-related occupational exposures and the use of PEP. Furthermore, unsafe practices are frequently observed, placing patients and healthcare workers at risk of infection.

knowledge and practice of PEP for HIV/HBV. As a result, the study recommended the establishment of PEP training centre with proper guidelines in order to enhance the utilization of PEP.

No empirical data exists on the knowledge and attitudes of HCWs toward post exposure prophylaxis following occupational exposure to the blood-borne viruses at Aswan University Hospital. Hence the study will apply interventions in the form of an education module designed to suit the need of each of these categories of HCWs (doctors, nurses, and ward aides). Furthermore, the study seeks to implement and evaluate the effectiveness of an education program regarding post exposure prophylaxis on their change in knowledge, attitude, and practice.

ELIGIBILITY:
Inclusion Criteria:

1. HCWs at the selected departments (physicians, nurses and housekeepers).
2. Age >18 years old and below 60 years old in both Genders.
3. HCWs which have direct contact with blood and body fluids.

Exclusion Criteria:

1. Age<18 years old and above 60 years old.
2. Non-medical staff at Aswan university hospital.
3. Health care workers which have no contact with blood or body fluids.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Health Practice Change | 3 Months
  Assessment of participants after taking health education lecturers about post-exposure prophylaxis regrading to knowledge, attitude and practice and this done by questionnaire as :The questionnaire consisted of three sections assessing knowledge, attitude, and practice regarding post-exposure prophylaxis (PEP).
  Section B assessed knowledge using nine close-ended questions, with adequate knowledge defined as ≥75% correct answers.
  Section C included seven items evaluating attitudes toward the importance and effectiveness of PEP, with scores ≥75% indicating a good attitude.
  Section D assessed PEP practices through nine questions, and good practice was defined as positive responses to more than 75% of items.

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa Sayed Abdelrheem, M.D, Study Chair — Associate Professor of Public Health and Community Medicine, Faculty of medicine, Aswan University
Locations (1):
- Aswan faculty of Medicine, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided